CLINICAL TRIAL: NCT02402725
Title: A Phase II, Open-label, Single Center Study of Ultra-High Dose Dexamethasone (UHDD) Administered Intravenously and Orally as Monotherapy for the Treatment of Relapsed Multiple Myeloma
Brief Title: A Open-label Study of Ultra-High Dose Dexamethasone for Relapsed Multiple Myeloma
Acronym: UltraDex
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: poor accrual
Sponsor: Boston Medical Center (Other)
Responsible Party: Principal Investigator, John Mark Sloan, Principal Investigator, Boston Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-33781; UltraDex (Other: Boston Medical Center)
Record Dates: First submitted 2015-03-09; First posted 2015-03-30 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2017-02

CONDITIONS: Multiple Myeloma
Keywords: Relapsed Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Dexamethasone; dexamethasone acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ultra-high dose dexamethasone (Experimental): Ultra-high dose dexamethasone administered intravenously and orally
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — (1 cycle = 28 days) D1: Dexamethasone 100mg IV; Dex 24mg PO every 6 hrs (begin immediately after IV dex) D2: Dex 24mg PO every 6 hrs D3: Dex 24mg PO every 6 hrs
  Other Names: Dexamethasone Acetate

SUMMARY:
This is a phase II, open label, single-center study of ultra-high dose dexamethasone administered intravenously and orally as monotherapy for the treatment of relapsed multiple myeloma. Dexamethasone has known anti-myeloma activity, and has been studied extensively both alone, and in combination with other agents, in the treatment of multiple myeloma.

This study implements an optimal 2-stage design. In Stage 1, 10 patients will be enrolled. Each patient will receive 100mg of intravenous dexamethasone once on Day 1, immediately followed by 24mg of oral (PO) dexamethasone every 6 hours for 3 days (Days 1-3) in a 28-day cycle. After 4 cycles, the patients will be evaluated for efficacy and safety. If 2 or more of the original 10 patients experience a CR, very good partial response (VGPR), or PR, an additional 20 patients will be enrolled in Stage 2. The enrollment for Stage 2 will occur after the completion of 4 cycles of ultra-high dose dexamethasone. If <2 patients experience a CR, VGPR, or PR, the study will be discontinued. Patients will be treated until progression, intolerable side effects, or death.

The purpose of the proposed phase II study is to determine the overall response rate, progression free survival, and tolerability of "ultra-high" dose dexamethasone.

DETAILED DESCRIPTION:
STUDY OBJECTIVES

Primary objective:

• Determine antitumor activity of ultrahigh dose dexamethasone (UHDD) as monotherapy in relapsed multiple myeloma.

Secondary objectives:

* Characterize the safety and tolerability of UHDD as monotherapy in patients with relapsed multiple myeloma.
* Determine the progression free survival amongst responders.
* Determine the subset of patients in whom UHDD can be used as monotherapy for treatment of relapsed multiple myeloma

STUDY ENDPOINTS

Primary endpoint: To determine the anti-tumor activity of UHDD as monotherapy in patients with relapsed multiple myeloma as measured by the International Myeloma Working Group (IMWG) response criteria:

* Change from baseline in M protein component.
* Objective response rate (complete response [CR] + partial response [PR]) assessed according to IMWG response criteria.
* Disease control rate (CR+PR+stable disease [SD]).

Secondary endpoints:

* Safety and tolerability of UHDD
* Progression free survival.
* Characteristics of patients responding to UHDD.

ELIGIBILITY:
Inclusion Criteria:

1. Relapsed multiple myeloma (MM) with measurable disease parameters according to the International Myeloma Working Group (IMWG) Criteria for the Diagnosis of Multiple Myeloma
2. Relapsed is defined as the development of disease progression following the achievement of stable disease (SD), partial response (PR), very good partial response (VGPR), complete response (CR) or stringent complete response (sCR) to the most recent anti-myeloma regimen
3. Received ≥ 2 prior regimen for MM
4. The patient or the patient's legal representative is able to understand the risks of the study and provide signed informed consent and authorization to use protected health information (in accordance with national and local privacy regulations)
5. ≥18 years of age
6. Karnofsky Performance Status score of ≥70
7. Able to adhere to the study visit schedule and other protocol requirements in the Investigator's opinion
8. Adequate hepatic function, as evidenced by serum bilirubin values <6.0 mg/dL and serum alanine transaminase (ALT) and/or aspartate transaminase (AST) values <3 × the upper limit of normal (ULN) of the local laboratory reference range. (Patients with isolated elevations in alkaline phosphatase [ALP] <5 × ULN in the presence of bony disease are not excluded from participating in the study)
9. If a female participant is of childbearing potential, she must have a negative pregnancy test (urine or serum) at baseline (Cycle 1, Day 0). (A female participant is considered to be NOT of childbearing potential if she has undergone bilateral oophorectomy or if she has been menopausal without a menstrual period for 12 consecutive months)

Exclusion Criteria:

1. Received any of the following therapies: Radiotherapy within 2 weeks of Cycle 1 Day 1; Systemic therapy within 3 weeks of Cycle 1 Day 1
2. Prior peripheral autologous stem cell transplant within 12 weeks of Cycle 1 Day 1
3. Prior allogeneic stem cell transplant
4. Active systemic infection requiring treatment
5. Active malignancy (the following are allowable: patients with basal cell carcinoma of the skin; superficial carcinoma of the bladder; carcinoma of the prostate with a current prostate-specific antigen <0.1 ng/mL; or cervical intraepithelial neoplasia).
6. Known or suspected human immunodeficiency virus (HIV) positive or hepatitis B surface antigen-positive status or is known or suspected to have an active hepatitis C infection
7. If female, patient is lactating
8. History of significant cardiovascular, neurological, endocrine, gastrointestinal, respiratory, or inflammatory illness that could preclude study participation, pose an undue medical hazard, or interfere with the interpretation of the study results, including, but not limited to, patients with:

   1. Congestive heart failure (New York Heart Association [NYHA] Class 3 or 4
   2. Unstable angina
   3. Cardiac arrhythmia
   4. Recent (within the preceding 6 months) myocardial infarction or stroke
   5. Hypertension requiring >3 medications for adequate control
   6. Chronic obstructive pulmonary disease
9. History of uncontrolled diabetes mellitus (Type I or II) (Hemoglobin A1C>8.5)
10. Any other medical, psychiatric, or social condition that would preclude participation in the study, pose an undue medical hazard, interfere with the conduct of the study, or interfere with interpretation of the study results
11. History of adverse reaction to dexamethasone or other corticosteroids.
12. History of allergic reaction attributable to any of the required prophylactic medications (proton pump inhibitor (PPI), fluconazole, trimethoprim-sulfamethoxazole) or reasonable alternative medications
13. Inability to monitor glucose at home with glucometer if glucose is found to be abnormal at any study center visit
14. Known or suspected AL Amyloidosis
15. Currently receiving an investigational agent for any reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-05; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Determine antitumor activity of ultrahigh dose dexamethasone (UHDD) as monotherapy in relapsed multiple myeloma. | 1 year

SECONDARY OUTCOMES:
Characterize the safety and tolerability by assessing the number of related adverse events of UHDD as monotherapy in patients with relapsed multiple myeloma. | 3 months
Determine the progression free survival amongst responders. | 5 years
Determine the subset of patients in whom UHDD can be used as monotherapy for treatment of relapsed multiple myeloma | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: John M Sloan, MD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No